CLINICAL TRIAL: NCT02767713
Title: The Role of Inflammatory and Stress Response in the Pathogenesis of Cognitive Dysfunction After Cardiac Surgery
Brief Title: Cognitive Dysfunction Following Cardiac Surgery
Acronym: CDCS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinical Hospital Center, Split (Other)
Responsible Party: Principal Investigator, Sandro Glumac, MD, Clinical Hospital Center, Split
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SPLIT1984
Record Dates: First submitted 2016-05-02; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Cognition Disorders; Cardiac Surgical Procedures; dexamethasone
MeSH Terms: conditions — Postoperative Cognitive Complications; Cognition Disorders | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone dose of 0.1 mg/kg was administered intravenously 10h before surgery
  Interventions: Drug: Dexamethasone
- Control (Placebo Comparator): Equal volume of normal saline (placebo) was administered intravenously 10h before surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Intravenous dexamethasone (0.1 mg/kg) was administered 10 hours before surgery.
  Other Names: Dexasone
  Arms: Dexamethasone
Other: Placebo — Normal saline (placebo) in the equal volume as active treatment was administered 10 hours before surgery.
  Other Names: Inactive substance
  Arms: Control

SUMMARY:
Postoperative cognitive dysfunction (POCD) is the most common complication after cardiac surgery. This prospective study was conducted to investigate the mechanisms of development of POCD following cardiac surgery taking into account surgical technique (with use or no use of extracorporeal circulation). The investigators focused on the role of inflammatory and stress response to surgical procedure as potential factors involved in the pathogenesis of cognitive dysfunction. Systematic inflammatory response in patients undergoing on-pump or off-pump surgery was analyzed by measuring serum levels of C reactive protein (CRP) and occurrence of systemic inflammatory response syndrome (SIRS). Stress response to surgery was evaluated following cortisol levels and its daily variations. The degree of cognitive dysfunction was assessed based on serum levels of S100β. The effect of dexamethasone on the levels of stress and inflammatory response biomarkers, serum levels of S100β, as well as on the development of POCD was compared with control group that received normal saline.

DETAILED DESCRIPTION:
This is a prospective, randomized, double blind, controlled trial. Following detailed past medical history assessment, two days before the surgical procedure neurocognitive function tests, depression and anxiety tests were carried out to assess the participants. Neurocognitive and anxiety tests were repeated on the 6th day after surgical procedure. A battery of tests lasting approximately 40 minutes were administered by a trained neuropsychologist from the Clinical Hospital Center, Split in a standardized fashion, at the same time of the day (10:00 AM) and in the same room at the Cardiac surgery ward. The investigators used a validated battery of tests which enabled the assessment of psychomotor speed, visual-motor coordination, concentration, attention, short-term memory and aspects of executive functioning. The evaluation was based on the following tests: Mini Mental State Examination (MMSE), Wechsler Memory Scale (WMS I & II), Trail Making Test (TMT A & B), Symbol Digit Modalities Test (SDMT), Controlled Oral Word Association Test (COWAT) and PsychE computer test. All of the tests except TMT A & B have alternate forms. Croatian versions of Beck Depression Inventory-Second Edition (BDI II) and State-Trait Anxiety Inventory (STAI-M) were used for preoperative depression and trait and state anxiety assessment, respectively.

One day before the surgery (08:00 AM) blood samples were collected for determination of levels of S100β protein, cortisol and other routine laboratory parameters (white blood cell count (WBC), hematocrit, creatinine, glucose, albumin, sodium, potassium, C reactive protein (CRP), Troponin I hs).

Participants were randomized into two groups to receive either intravenous dexamethasone 0.1 mg/kg or the same volume of normal saline i.v. 10 hours before the surgery. Random sequence generator was used to determine participant allocation.

Anesthesia in all patients was based on fentanyl, midazolam, vecuronium and sevoflurane. The depth of anesthesia was monitored using bispectral index (BIS). During cardiopulmonary bypass alpha-stat technique was used with the maintenance of normothermia (35.5-36.5°C) or spontaneous hypothermia (up to 32°C). With the off-pump technique, the core temperature was maintained between 36 and 37°C. Surgical technique was standardized. Routine hemodynamic monitoring was performed throughout the surgery and continued on the first postoperative day. Plasma levels of S100β protein were determined 6 h and 30 h following the end of on-pump surgery, and 3 h following the end of off-pump surgery. C reactive protein levels and other routine laboratory parameters were measured from blood samples collected 1 h, 4 h and 12 h postoperatively. On the first postoperative day blood samples were collected at 08:00 AM to determine cortisol levels, C reactive protein and other routine laboratory parameters, and cortisol was also measured on the same day at 04:00 PM, and 12:00 AM. C reactive protein and other routine laboratory parameters were repeatedly measured at 08:00 AM on the following postoperative days, except for cortisol levels which were measured on postoperative days 3 and 5. Registered nurse carried out the standardized test (Delirium Observation Screening Scale (DOS) scale) to assess the patients for the development of postoperative delirium from second to fifth postoperative day (at 07:00 AM, 02:00 PM and 10:00 PM).

ELIGIBILITY:
Inclusion Criteria:

* Participants undergoing cardiac surgery: coronary artery bypass grafting, heart valve surgery or a combined procedure,
* Procedure must be elective

Exclusion Criteria:

* Symptomatic cerebrovascular disease,
* Cerebrovascular incident in last 3 years,
* Neurodegenerative disease,
* Psychiatric disease,
* Visual, hearing or motor impairment interfering with cognitive testing,
* Carotid artery stenosis ( ≥50%),
* Myocardial infarction within last 3 months,
* Left ventricular ejection fraction of ≤35%,
* Previous cardiac or carotid surgery,
* Uncontrolled systemic hypertension (blood pressure≥180/110 mmHg),
* Corticosteroid-dependent asthma,
* Chronic obstructive pulmonary disease (COPD),
* Malignancy, liver disease (aspartate transaminase (AST), alanine transaminase (ALT) or bilirubin ˃1.5x above reference range),
* Kidney disease (serum creatinine ˃1.7 mg/dl or blood urea nitrogen ˃50 mg/dL),
* Uncontrolled diabetes mellitus (postprandial glucose ˃200 mg/dL or hemoglobin A1c ˃9%),
* Endocrine and metabolic diseases, requiring steroid treatment longer than 7 days in the past year,
* Alcohol or controlled substance abuse,
* Individuals without primary school education,
* Preoperative C reactive protein ˃0.5 mg/dL,
* Preoperative white blood cell count <3 x109/L or ˃11 x109/L,
* Preoperative Mini mental score <26 points,
* Preoperative Beck's depression inventory score ˃ 19 points,
* Intraoperative plan change (conversion from "off-pump" to "on-pump" and vice versa),
* Need for deep hypothermic circulatory arrest,
* Additional corticosteroid treatment throughout the study period.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Difference in occurrence of postoperative cognitive dysfunction between control and intervention group at six days after surgery as determined by using a validated battery of cognitive tests | 9 days
  Difference in occurrence of postoperative cognitive dysfunction between control and intervention group at sixth postoperative day as determined by using a validated battery of cognitive tests that assess global cognitive function, psychomotor speed, visual-motor coordination, concentration, attention, short-term memory, learning curve and aspects of executive functioning. Time points of assessment are two days before surgery and six days after surgery in both study arms.

SECONDARY OUTCOMES:
Change in serum levels of S100β protein from baseline to first postoperative day | 3 days
  Serum levels of S100β protein were determined the day before surgery at 08:00 AM; 6 h and 30 h following the end of on-pump surgery; and 3 h following the end of off-pump surgery.
Difference in S100β serum protein levels between control and intervention group on the day of surgery and first postoperative day | 7 days
Change in serum cortisol levels from baseline to fifth postoperative day | 7 days
  Cortisol levels were determined on the day before surgery at 08:00 AM; on the first postoperative day at 08:00 AM, 04:00 PM, and 12:00 AM; and at 08:00 AM on the third and fifth postoperative days.
Difference in serum cortisol levels between control and intervention group on the first, third and fifth postoperative days | 7 days
Change in serum C reactive protein levels from baseline to fifth postoperative day | 7 days
  Baseline CRP levels were determined on the day before surgery at 08:00 AM, 1 h, 4 h and 12 h postoperatively; and at 08:00 AM from the first until fifth postoperative day.
Difference in serum C reactive protein levels between control and intervention group on the day of surgery until the fifth postoperative day | 7 days
Difference in occurrence of systemic inflammatory response syndrome between control and intervention group within 48 h after surgery as determined by measuring body temperature, heart rate, respiratory rate, and white blood cell count. | 48 hours
Difference in occurrence of postoperative delirium between control and intervention group as determined from second until sixth postoperative day by using Delirium Observation Screening Scale | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Nenad Karanovic, MD, PhD, Study Director — Clinical Hospital Center, Split

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ottens TH, Dieleman JM, Sauer AM, Peelen LM, Nierich AP, de Groot WJ, Nathoe HM, Buijsrogge MP, Kalkman CJ, van Dijk D; DExamethasone for Cardiac Surgery (DECS) Study Group. Effects of dexamethasone on cognitive decline after cardiac surgery: a randomized clinical trial. Anesthesiology. 2014 Sep;121(3):492-500. doi: 10.1097/ALN.0000000000000336. PMID 25225745
- [Background] Newman MF, Kirchner JL, Phillips-Bute B, Gaver V, Grocott H, Jones RH, Mark DB, Reves JG, Blumenthal JA; Neurological Outcome Research Group and the Cardiothoracic Anesthesiology Research Endeavors Investigators. Longitudinal assessment of neurocognitive function after coronary-artery bypass surgery. N Engl J Med. 2001 Feb 8;344(6):395-402. doi: 10.1056/NEJM200102083440601. PMID 11172175
- [Background] Roach GW, Kanchuger M, Mangano CM, Newman M, Nussmeier N, Wolman R, Aggarwal A, Marschall K, Graham SH, Ley C. Adverse cerebral outcomes after coronary bypass surgery. Multicenter Study of Perioperative Ischemia Research Group and the Ischemia Research and Education Foundation Investigators. N Engl J Med. 1996 Dec 19;335(25):1857-63. doi: 10.1056/NEJM199612193352501. PMID 8948560
- [Background] Hudetz JA, Gandhi SD, Iqbal Z, Patterson KM, Pagel PS. Elevated postoperative inflammatory biomarkers are associated with short- and medium-term cognitive dysfunction after coronary artery surgery. J Anesth. 2011 Feb;25(1):1-9. doi: 10.1007/s00540-010-1042-y. PMID 21061037
- [Background] Rasmussen LS, O'Brien JT, Silverstein JH, Johnson TW, Siersma VD, Canet J, Jolles J, Hanning CD, Kuipers HM, Abildstrom H, Papaioannou A, Raeder J, Yli-Hankala A, Sneyd JR, Munoz L, Moller JT; ISPOCD2 Investigators. Is peri-operative cortisol secretion related to post-operative cognitive dysfunction? Acta Anaesthesiol Scand. 2005 Oct;49(9):1225-31. doi: 10.1111/j.1399-6576.2005.00791.x. PMID 16146456
- [Background] Mu DL, Li LH, Wang DX, Li N, Shan GJ, Li J, Yu QJ, Shi CX. High postoperative serum cortisol level is associated with increased risk of cognitive dysfunction early after coronary artery bypass graft surgery: a prospective cohort study. PLoS One. 2013 Oct 15;8(10):e77637. doi: 10.1371/journal.pone.0077637. eCollection 2013. PMID 24143249
- [Background] Phillips-Bute B, Mathew JP, Blumenthal JA, Grocott HP, Laskowitz DT, Jones RH, Mark DB, Newman MF. Association of neurocognitive function and quality of life 1 year after coronary artery bypass graft (CABG) surgery. Psychosom Med. 2006 May-Jun;68(3):369-75. doi: 10.1097/01.psy.0000221272.77984.e2. PMID 16738066
- [Background] Jensen BO, Hughes P, Rasmussen LS, Pedersen PU, Steinbruchel DA. Cognitive outcomes in elderly high-risk patients after off-pump versus conventional coronary artery bypass grafting: a randomized trial. Circulation. 2006 Jun 20;113(24):2790-5. doi: 10.1161/CIRCULATIONAHA.105.587931. Epub 2006 Jun 12. PMID 16769915
- [Background] Parolari A, Camera M, Alamanni F, Naliato M, Polvani GL, Agrifoglio M, Brambilla M, Biancardi C, Mussoni L, Biglioli P, Tremoli E. Systemic inflammation after on-pump and off-pump coronary bypass surgery: a one-month follow-up. Ann Thorac Surg. 2007 Sep;84(3):823-8. doi: 10.1016/j.athoracsur.2007.04.048. PMID 17720383
- [Background] Canet J, Raeder J, Rasmussen LS, Enlund M, Kuipers HM, Hanning CD, Jolles J, Korttila K, Siersma VD, Dodds C, Abildstrom H, Sneyd JR, Vila P, Johnson T, Munoz Corsini L, Silverstein JH, Nielsen IK, Moller JT; ISPOCD2 investigators. Cognitive dysfunction after minor surgery in the elderly. Acta Anaesthesiol Scand. 2003 Nov;47(10):1204-10. doi: 10.1046/j.1399-6576.2003.00238.x. PMID 14616316
- [Background] Ernest CS, Worcester MU, Tatoulis J, Elliott PC, Murphy BM, Higgins RO, Le Grande MR, Goble AJ. Neurocognitive outcomes in off-pump versus on-pump bypass surgery: a randomized controlled trial. Ann Thorac Surg. 2006 Jun;81(6):2105-14. doi: 10.1016/j.athoracsur.2006.01.008. PMID 16731138
- [Derived] Glumac S, Kardum G, Sodic L, Bulat C, Covic I, Carev M, Karanovic N. Longitudinal assessment of preoperative dexamethasone administration on cognitive function after cardiac surgery: a 4-year follow-up of a randomized controlled trial. BMC Anesthesiol. 2021 Apr 23;21(1):129. doi: 10.1186/s12871-021-01348-z. PMID 33892653
- [Derived] Glumac S, Kardum G, Sodic L, Supe-Domic D, Karanovic N. Effects of dexamethasone on early cognitive decline after cardiac surgery: A randomised controlled trial. Eur J Anaesthesiol. 2017 Nov;34(11):776-784. doi: 10.1097/EJA.0000000000000647. PMID 28985195